CLINICAL TRIAL: NCT01591837
Title: A Phase IV, Single-Centre, Open-label Study to Evaluate the Immunogenicity and Safety of the 2012/2013 Formulation of the Enzira® Vaccine in Two Groups of Healthy Volunteers: 'Adults' (Aged 18 to 59 Years) and 'Older Adults' (Aged 60 Years or Older)
Brief Title: A Study to Assess the Immunogenicity and Safety of CSL's 2012/2013 Formulation of Enzira® Vaccine in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CSLCT-ASU-12-76; 2012-001101-24 (EudraCT Number)
Record Dates: First submitted 2012-05-03; First posted 2012-05-04 (Estimated); Results first posted 2013-11-18 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-04

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human

ARMS (2):
- Adults (Experimental): Healthy volunteers aged 18 to 59 years received a single 0.5 mL dose of CSL Influenza Vaccine by intramuscular or subcutaneous injection.
  Interventions: Biological: CSL Influenza Vaccine
- Older Adults (Experimental): Healthy volunteers aged 60 years or older received a single 0.5 mL dose of CSL Influenza Vaccine by intramuscular or subcutaneous injection.
  Interventions: Biological: CSL Influenza Vaccine

INTERVENTIONS:
Biological: CSL Influenza Vaccine — The study vaccine (CSL Influenza Vaccine) is a sterile, thiomersal-free suspension containing 45 mcg total haemagglutinin antigen per 0.5 mL dose (15 mcg each of the three recommended influenza strains for the Northern Hemisphere 2012/2013 influenza season). The vaccine will be administered by intramuscular or subcutaneous injection.
  Other Names: Enzira® vaccine; Afluria® vaccine

SUMMARY:
This is a study to assess the immune (antibody) response and safety of the 2012/2013 formulation of Enzira® (CSL Influenza vaccine) in healthy adult volunteers aged 18 years or older.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 years or older at the time of vaccination.
* Females of child-bearing potential (i.e., ovulating, pre-menopausal, not surgically sterile) must be abstinent or be willing to use a medically accepted contraceptive regimen for the duration of the study. Females of child-bearing potential must return a negative urine pregnancy test result prior to vaccination with the vaccine.

Exclusion Criteria:

* Known hypersensitivity to a previous vaccination with influenza vaccine or allergy to eggs, ovalbumin, chicken protein, neomycin, polymyxin, or any components of the vaccine.
* Clinical signs of an active infection.
* A clinically significant medical condition.
* Vaccination with a seasonal or experimental influenza virus vaccine in the 6 months preceding study entry.
* Females who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Director Vaccines, Study Director — Seqirus
Locations (1):
- Study Site, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adults | Older Adults
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adults | Older Adults | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (12.50) | 69.2 (6.69) | 52.2 (19.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 29 | 67
  Male | 22 | 31 | 53

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Evaluable Participants Achieving Seroconversion or Significant Increase in Antibody Titre.
Description: As per the criteria specified in the CPMP/BWP/214/96 Note for Guidance on Harmonisation of Requirements for Influenza Vaccines. For haemagglutination inhibition (HI), seroconversion (H1N1, H3N2, and B influenza virus strains) was defined as achieving a post-vaccination titre of ≥ 40 for those participants with a pre-vaccination HI titre of < 10. A significant increase (H1N1, H3N2, and B influenza virus strains) was defined as a four-fold or greater increase in HI titre for those participants with a pre-vaccination HI titre of ≥ 10.
Time Frame: Approximately 21 days after vaccination
Population: The Evaluable Population included all participants who were vaccinated with CSL Influenza Vaccine, provided both pre- and post-vaccination antibody titer results, did not use a prohibited medication as per the protocol, and were not excluded from the analysis according to the elimination criteria.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adults | Older Adults
Number analyzed (Participants) | 59 | 59
percentage of participants
  H1N1 strain | 79.7 [67.2 to 89.0] | 55.9 [42.4 to 68.8]
  H3N2 strain | 86.4 [75.0 to 94.0] | 64.4 [50.9 to 76.4]
  B strain | 59.3 [45.7 to 71.9] | 18.6 [9.7 to 30.9]

2. Primary Outcome: The Geometric Mean Fold Increase (GMFI) in Antibody Titre After Vaccination.
Description: GMFI (H1N1, H3N2, and B influenza virus strains) was defined as the geometric mean of the fold increases of post-vaccination antibody titre over the pre-vaccination antibody titre.
Time Frame: Approximately 21 days after vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean fold increase
Arm/Group | Adults | Older Adults
Number analyzed (Participants) | 59 | 59
geometric mean fold increase
  H1N1 strain | 17.51 [11.857 to 25.852] | 7.78 [5.217 to 11.614]
  H3N2 strain | 21.80 [14.332 to 33.164] | 9.88 [6.316 to 15.468]
  B strain | 7.34 [5.592 to 9.634] | 2.44 [1.913 to 3.118]

3. Primary Outcome: The Percentage of Evaluable Participants Achieving a HI Titre ≥ 40 or Single Radial Haemolysis (SRH) Area ≥ 25 mm2.
Description: For the H1N1, H3N2, and B influenza virus strains. Note: No SRH data were collected.
Time Frame: Approximately 21 days after vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adults | Older Adults
Number analyzed (Participants) | 59 | 59
percentage of participants
  H1N1 strain | 94.9 [85.9 to 98.9] | 84.7 [73.0 to 92.8]
  H3N2 strain | 100.0 [93.9 to 100.0] | 100.0 [93.9 to 100.0]
  B strain | 66.1 [52.6 to 77.9] | 18.6 [9.7 to 30.9]

4. Secondary Outcome: Frequency and Intensity of Any Solicited Adverse Events (AEs).
Description: The percentage of participants reporting any solicited AEs and the percentage of participants reporting any solicited AEs with severe intensity. Note: Intensity of solicited AEs was collected for temperature only.
  Solicited local AEs collected included induration >50 mm, erythema, ecchymosis, and pain at the vaccination site.
  Solicited systemic AEs collected included temperature above 38.0°C, chills, and malaise.
  Solicited AE intensity grading: Mild: symptoms were easily tolerated and there was no interference with daily activities; Moderate: enough discomfort to cause some interference with daily activities; Severe: symptoms that prevented normal, everyday activities.
Time Frame: During the 4 days after vaccination (Day 0 plus 3 days)
Population: The Safety Population included all participants who received CSL Influenza Vaccine and provided follow-up safety data.
Measure: Number; unit: percentage of participants
Arm/Group | Adults | Older Adults
Number analyzed (Participants) | 60 | 60
percentage of participants
  Any solicited local AE | 46.7 | 18.3
  Induration > 50 mm | 0.0 | 3.3
  Erythema | 15.0 | 6.7
  Ecchymosis | 6.7 | 3.3
  Pain | 41.7 | 10.0
  Any solicited systemic AE | 15.0 | 6.7
  Temperature > 38°C for ≥ 24 hours | 0 | 1.7
  Severe temperature (> 40°C) | 0 | 1.7
  Chills | 10.0 | 3.3
  Malaise | 13.3 | 6.7

5. Secondary Outcome: Frequency of Any Unsolicited AEs.
Description: The percentage of participants reporting any unsolicited AEs. Unsolicited AEs included AEs other than those specifically solicited.
Time Frame: After vaccination until the end of the study; approximately 21 days
Population: The Safety Population included all participants who received CSL Influenza Vaccine and provided follow-up safety data.
Measure: Number; unit: percentage of participants
Arm/Group | Adults | Older Adults
Number analyzed (Participants) | 60 | 60
percentage of participants | 53.3 | 36.7

ADVERSE EVENTS:
Time Frame: For solicited AEs: During the 4 days after vaccination (Day 0 plus 3 days); For unsolicited AEs and serious AEs (SAEs): After vaccination until the end of the study (approximately 21 days).
Description: The other AEs presented include solicited and unsolicited AEs.
  The Safety Population included all participants who received CSL Influenza Vaccine and provided follow-up safety data.
Arm/Group | Adults | Older Adults
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 36/60 | 18/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adults (N=60) | Older Adults (N=60)
Pain (General disorders) | 25 (26) | 6 (6)
Erythema (General disorders) | 9 (9) | 4 (4)
Ecchymosis (General disorders) | 4 (4) | 2 (2)
Malaise (General disorders) | 8 (9) | 4 (5)
Chills (General disorders) | 6 (6) | 2 (2)
Headache (Nervous system disorders) | 15 (17) | 5 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 5 (5)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSL agreements and restrictions on publishing may vary with individual investigators; however, CSL will not prohibit any investigator from publishing. CSL supports the publication of results from all centers of a multi-center trial and generally requires that reports based on single-site data not precede the primary publication of the entire clinical trial.